CLINICAL TRIAL: NCT01657617
Title: Stereotactic Body Radiation Therapy for Post-chemoradiation Residual Disease in Stage II/III Non-small Cell Lung Cancer
Brief Title: Stereotactic Body Radiation Therapy in Stage II/III Non Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ronald McGarry (Other)
Responsible Party: Sponsor-Investigator, Ronald McGarry, Professor, Radiation Medicine, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-07-RAD-01
Record Dates: First submitted 2012-01-17; First posted 2012-08-06 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiation Therapy (Experimental): Boost Stereotactic Body Radiation Therapy (SBRT)
  Interventions: Radiation: Boost Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Boost Stereotactic Body Radiation Therapy — The dose and fractionation scheme utilized will be based on the location of the patient's residual disease. For patients with:
  Peripheral Tumors: Treatment will consist of 2 fractions of radiation, with a minimum of 40 hours separating each fraction. Two fractions of 10 Gy with inhomogeneity correction will be delivered to the prescription line at the edge of the PTV for a total of 20 Gy. This will yield a total BED of 110 Gy.
  Medial Tumors: Treatment will consist of 3 fractions of radiation, with a minimum of 40 hours separating each fraction. Three fractions of 6.5 Gy with inhomogeneity correction will be delivered to the prescription line at the edge of the PTV for a total of 19.5 Gy. This will yield a total BED 102.2 Gy.

SUMMARY:
It is apparent that local control for Non-small Cell Lung Cancer (NSCLC) remains a significant problem. Conventional radiation therapy techniques have limitations for the dose that can be delivered to a chest tumor mass due to the adjacent dose limiting organs. Mounting evidence supports the use of hypofractionated stereotactically delivered radiation therapy to control lung cancer with acceptable toxicity profiles.

Thus the investigators propose to increase the doses of radiation to residual masses of NSCL to a BED > 100 Gy by the addition of two fractions of stereotactically delivered boost radiation therapy to residual disease post-conventional chemoradiation to at least 59.4 Gy in 180 cGy fractions. Using the linear quadratic equation to model doses of radiation therapy, 59.4 Gy would have a BED of approximately 70 Gy. Single fraction stereotactic body radiation therapy (SBRT) of 10 Gy would have a BED of approximately 20 Gy. Thus the addition of two fractions of 10Gy of SBRT to limited volumes of PET residual disease would theoretically result in higher degrees of local control of lung cancer masses, achieving a minimum cumulative BED of approximately 110Gy-equivalent.

DETAILED DESCRIPTION:
Lung cancer represents one of the most challenging malignancies to manage. Cure rates have only marginally improved in the last 20 years. It is the most commonly fatal cancer in both men and women with overall 5 year survivals of 15%. Lung cancer kills more Americans than the next three most common malignancies combined.

Most non small cell lung cancer (NSCLC) presents at advanced stages. Only approximately 25% present with stage I/II disease, 40% with stage III and 35% patients present with stage IV. (1) The optimal treatment of stage II/III NSCLC is complex. For those patients who are surgical candidates and a complete resection is technically feasible, radical surgery remains the standard of care. Traditionally, those patients with multiple N2 nodal levels or T4 disease are considered inoperable. Given that the average age of patients diagnosed with NSCLC is in their mid-60's and usually have long smoking histories, many patients are medically inoperable.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of non-small cell lung cancer (squamous cell carcinoma, adenocarcinoma, large cell carcinoma, bronchoalveolar cell carcinoma, or non-small cell carcinoma NOS) by either biopsy or cytology.
2. Clinical AJCC stage IIA (T1N1M0), IIB (T2,N1M0, T3,N0,M0) or IIIA (T1-3, N1-2,M0)/selected IIIB. In all cases, patients may be included at the discretion of the treating radiation oncologist if it will be likely the disease can be encompassed by the stereotactic boost will be included.
3. Patients with non-bulky (< 2.0-3.0 cm) hilar or mediastinal lymphadenopathy determined by pre-treatment CT scan, PET or mediastinoscopy
4. Must have completed a standard course of chemoradiation in accordance with NCCN Guidelines
5. One month following definitive chemoradiation, CT or PET-CT revealing limited volume residual disease within the site of primary tumour mass (post-chemo/RT mass </= 7.0 cm). Patients with a CR and no obvious target are not eligible.
6. must be able to fit into the Elekta Stereotactic body frame
7. Patients must be ≥ 18 years of age.
8. The patient's ECOG performance status must be 0-2.
9. Women of childbearing potential and male participants must use an effective contraceptive method.
10. Patients must sign a study-specific consent form.

Exclusion Criteria:

1. Any other active cancer OR No prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or other cancer from which the patient has been disease-free for 5 years.
2. Patients with other systemic illness, or have not recovered adequately from their primary treatment or who have evidence of progression of their lung cancer prior to therapy that, in the investigators opinions, would preclude their inclusion
3. Plans for the patient to receive other concomitant antineoplastic therapy while on this protocol, except at disease progression. Patients may be allowed to use bisphosphonates for hypercalcemia.
4. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-10-01 (Actual); Primary Completion 2014-06-05 (Actual); Study Completion 2018-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald C. McGarry, MD, PhD., Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the oncology clinics at the University of Kentucky between 2007 and 2014
Groups:
- Radiation Therapy: Boost Stereotactic Body Radiation Therapy
  Boost Stereotactic Body Radiation Therapy: The dose and fractionation scheme utilized will be based on the location of the patient's residual disease. For patients with:
  Peripheral Tumors: Treatment will consist of 2 fractions of radiation, with a minimum of 40 hours separating each fraction. Two fractions of 10 Gy with inhomogeneity correction will be delivered to the prescription line at the edge of the PTV for a total of 20 Gy. This will yield a total BED of 110 Gy.
  Medial Tumors: Treatment will consist of 3 fractions of radiation, with a minimum of 40 hours separating each fraction. Three fractions of 6.5 Gy with inhomogeneity correction will be delivered to the prescription line at the edge of the PTV for a total of 19.5 Gy. This will yield a total BED 102.2 Gy.
Period: Overall Study
Arm/Group | Radiation Therapy
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 63 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 31
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Boost Dose Toxicity
Description: Pneumonitis will be used as a marker of lung toxicity as a result of the Boost treatment. Participants will follow up with their treating physician annually for five years after treatment with SBRT . Any incidence of pneumonitis will be documented. Data will be presented as the percent of subjects receiving SBRT that required treatment for pneumonitis.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 35
Participants | 5

2. Secondary Outcome: Primary Tumor Relapse Following SBRT
Description: The response rates of the residual primary tumor following SBRT boost will be determined using a modified version of the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Data will be presented as the percent of participants with recurrence of the primary tumor after extended follow up, up to 5 years.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 35
Participants | 8

ADVERSE EVENTS:
Arm/Group | Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 30/35
Serious Adverse Events (participants affected / at risk) | 2/35
Other Adverse Events (participants affected / at risk) | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy (N=35)
Fatal hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This study was a single site, low enrollment proof of concept trial of the effectiveness of local radiation following SOC chemotherapy. The data are promising; however, larger trials are in order to demonstrate its full therapeutic value.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-07-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT01657617/Prot_SAP_000.pdf